CLINICAL TRIAL: NCT06470529
Title: Comparative Evaluation of Incidence of Cardiovascular Events Among Different Drug-Eluting Stent Types
Brief Title: MACE in Different Drug-Eluting Stents
Status: Completed | Type: Observational
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Other Study IDs: IR.SUMS.MED.RED.1402.409
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease; Stent Restenosis
Keywords: Percutaneous coronary intervention; Major adverse coronary events (MACE); drug eluting stents
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCI: Post PCI patients with drug eluting stents
  Interventions: Device: drug eluting stents

INTERVENTIONS:
Device: drug eluting stents — different types of drug eluting stents

SUMMARY:
In this retrospective cohort study, all patients from Iranian registry were recruited and follow up after 5 years were recorded for MACE, and its relation to type and demographic data were evaluated

DETAILED DESCRIPTION:
This retrospective cohort study involved 4,438 individuals who received a PCI from March 2019 to February 2021. Data was obtained from the Iranian Network of Cardiovascular Research Registry ( which registered post PCI patients all around Iran in more than 40 public and private hospitals) and the database of Professor Kojuri Cardiology Clinic (Niyayesh St., Shiraz, Iran, www.kojuriclinic.com). After each procedure, expert cardiologists recorded baseline demographic data, prior medical history, angiography, and angioplasty reports.

Demographic data such as age, gender, body mass index (BMI), family history of CAD, prior CAD history, hypertension (HTN), diabetes mellitus (DM), hyperlipidemia (HLP), and kidney diseases were obtained from the database. Data on the prevalence of cigarette smoking, opium addiction, and alcohol addiction were collected. Additionally, information on clinical manifestations of the disease, including stable angina, unstable angina, ST-elevation myocardial infarction (STEMI), and non-ST elevation myocardial infarction (NSTEMI), was extracted.

According to the American Heart Association (AHA), stage 1 hypertension is defined as a systolic blood pressure of 130-139 mmHg or diastolic blood pressure of 80-89 mmHg ; Hypertension was defined as stage 1 or higher blood pressure. DM was defined according to The American Diabetes Association as having a hemoglobin A1c level of at least 6.5%, a fasting plasma glucose (FPG) level of 126 mg/dl or higher, an oral glucose tolerance test (OGTT) level of 200 mg/dl or greater, or a random plasma glucose level of 200 mg/dl or above . For defining dyslipidemia, based on the 2019 AHA guideline, a low-density lipoprotein cholesterol (LDL-C) level exceeding 160 mg/dl or a non-high-density lipoprotein cholesterol (non-HDL-C) over 190 mg/dl were considered . Individuals with ≤1 month of smoking cessation were considered current smokers .

Angiography and angioplasty data Angiography and angioplasty data were gathered, including the type and location of coronary artery lesions and the type, location, size, diameter, and number of stents. Drug-eluting stents encompass a variety of types, notably the biolimus-eluting stent (BES), amphilimus-eluting stent (AES), SES, ZES, PES, and EES. Within the BES category, a notable example is the BioMatrix™ stent, while SES includes options like BioMimeTM, Orsiro®, Cre8, SUPRAFLEX, ULTIMASTERTM, and Coroflex® ISAR. ZES variants include the Resolute Onyx™ and Resolute Integrity™ stents, whereas EES comprises options such as Promus PREMIER, Promus Element™, and XIENCE™. Polymer-coated drug-eluting stents (PC-DES) include BioMatrix™, BioMimeTM, Orsiro®, SUPRAFLEX, ULTIMASTERTM, Resolute Onyx™, Resolute Integrity™, Promus PREMIER, Promus Element™, and XIENCE™. Conversely, polymer-free drug-eluting stents (PF-DES) are exemplified by Cre8 and Coroflex® ISAR. Regarding generational classification, the first generation includes BioMimeTM, Orsiro®, Cre8, SUPRAFLEX, ULTIMASTERTM, and Coroflex® ISAR. Notable second-generation members are Promus PREMIER, Promus Element, and XIENCE™, alongside Resolute Onyx™ and Resolute Integrity™. Finally, the BioMatrix™ stent represents the third generation.

Data of ballooning, including predilatation, postdilatation, and the number of balloons used were collected. Different angioplasty techniques, including kissing and overlapping were collected .Coronary legions were classified according to the ACC/AHA classification: type A: <10 mm, non-angulated, smooth, little calcification, not totally occlusive, not ostial, no major branch involvement, no thrombus; type B: 10-20 mm, eccentric, moderately tortuous, 45-90º, irregular, moderate to heavy calcification, ostial, bifurcation lesions, some thrombus (subcategories: B1: one characteristic; B2: two or more characteristics), and type C: diffuse, extremely angulated, >90º, inability to protect major side branch, degenerated vein graft .

Follow-up Patients were contacted by phone to explain the study plans and obtain informed consent. They were asked about MACEs occurring within two years following angioplasty, which includes myocardial infarction, acute heart failure, stroke, and death from cardiac diseases, as well as any revascularization. Additionally, the date of MACE occurrence after angioplasty was recorded, and information on non-cardiac-related deaths was collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary angioplasty who received at least one type of DES

Exclusion Criteria:

* Patients who received multiple types of stents
* Patients who need emergency operation post PCI

Ages: 36 Years to 82 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients all around the Iran, from 40 hospitals, who undergone PCI as elective or emergency patients
Sampling Method: Non-Probability Sample
Enrollment: 4159 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Major adverse coronary events | 5 years
  Total sum of Myocardial infarction (MI), Hospital admission, Death, reoperation or re PCI,

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No
Data was available based on rational request